CLINICAL TRIAL: NCT04262492
Title: OBServaToire INternational Des Patients AnTiphospholipidEs traités Par Anticoagulants Oraux Directs
Brief Title: International Registry of Thrombotic APS Patients Treated With Direct Oral Anticoagulants
Acronym: OBSTINATE
Status: Recruiting | Type: Observational
Sponsor: Stéphane Zuily (Other)
Collaborators: International Society on Thrombosis and Haemostasis (Unknown)
Responsible Party: Sponsor-Investigator, Stéphane Zuily, Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2019-A01415-52
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Antiphospholipid Syndrome; Thrombosis; Anticoagulants Causing Adverse Effects in Therapeutic Use
Keywords: antiphospholipid syndrome; direct oral anticoagulants
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombosis | interventions — Rivaroxaban; Dabigatran; apixaban; edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 10 mg or 15 mg or 20 mg OD Dabigatran 110 mg or 150 mg BID Apixaban 2.5 mg or 5 mg or 10 mg BID
  Other Names: Dabigatran; Apixaban; Edoxaban

SUMMARY:
This registry, currently being established will ensure consistency of data collection and provide safety information in non high-risk APS patients currently on DOACs.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving a comprehensive information about the study, and not opposed to participate
* Age ≥ 18 yo
* Classification of definite APS according to revised Sapporo-Sydney criteria
* Direct oral anticoagulant treatment prescribed during at least 6 months or with the possibility of follow-up of at least 6 months

Exclusion Criteria:

* Incomplete revised Sapporo-Sydney criteria
* No data regarding the recurrent thrombosis
* Pregnant woman
* Age < 18 yo

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Thrombotic APS patients according to revised Sapporo-Sydney criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Recurrent Thrombosis | 6 months
  Rate of Recurrent Thrombosis either arterial, venous or microvascular confirmed by a relevant exam

SECONDARY OUTCOMES:
Rate of Bleeding | 6 months
  Rate of Bleeding either severe or major or clinically relevant non-major bleeding according to ISTH classification
Rate of Non-Criteria Manifestations | 6 months
  Rate of Non-Criteria Manifestations according to Sydney criteria
Adherence to treatment | 6 months
  Rate of patients who have a good adherence to oral anticoagulants assessed by the Girerd questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Stéphane Zuily, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dufrost V, Risse J, Reshetnyak T, Satybaldyeva M, Du Y, Yan XX, Salta S, Gerotziafas G, Jing ZC, Elalamy I, Wahl D, Zuily S. Increased risk of thrombosis in antiphospholipid syndrome patients treated with direct oral anticoagulants. Results from an international patient-level data meta-analysis. Autoimmun Rev. 2018 Oct;17(10):1011-1021. doi: 10.1016/j.autrev.2018.04.009. Epub 2018 Aug 11. PMID 30103045
- [Background] Dufrost V, Risse J, Wahl D, Zuily S. Direct Oral Anticoagulants Use in Antiphospholipid Syndrome: Are These Drugs an Effective and Safe Alternative to Warfarin? A Systematic Review of the Literature: Response to Comment. Curr Rheumatol Rep. 2017 Aug;19(8):52. doi: 10.1007/s11926-017-0676-2. No abstract available. PMID 28741234
- See also: ISTH SSC LA/aPL project — https://cdn.ymaws.com/www.isth.org/resource/resmgr/subcommittees/registry_on_doacs_in_aps_pro.pdf
- See also: OBSTINATE webpage — https://apsnancy.com/Research-Projects.php